CLINICAL TRIAL: NCT02366455
Title: Knowing the Right Upper Lobe Anatomy Allows for the Efficient Use of the Right-sided Double Lumen Endobronchial Tube
Brief Title: New Measures for Tracheobronchial Anatomy
Acronym: ATB
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Jean Bussières, Anesthesiologist, Laval University
Other Study IDs: IUCPQ-ATB2014
Record Dates: First submitted 2015-02-12; First posted 2015-02-19 (Estimated); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Thoracic CT-scan; Right Upper Lobe Anatomy; Right Sided Double Lumen Endobronchial Tube

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thoracic CT-Scan: Measurement of the length of the right main stem bronchus and of the right upper lobe bronchus antero-posterior angulation on consecutive thoracic CT-Scan reconstruction
  Interventions: Procedure: Measurement of the length of the right main stem bronchus; Procedure: Measurement of the right upper lobe bronchus antero-posterior angulation

INTERVENTIONS:
Procedure: Measurement of the length of the right main stem bronchus — Measurement of the length of the right main stem bronchus on CT-Scan
Procedure: Measurement of the right upper lobe bronchus antero-posterior angulation — Measurement of the right upper lobe bronchus antero-posterior angulation on CT-Scan

SUMMARY:
The right-sided double lumen endobronchial tube (R-DLT) is seldom. The principal cause of reticence for using the R-DLT are the difficult positioning of its lateral orifice in front of the origin of the right upper lobe (RUL) and the variability of the length of the right main stem bronchus (RMSB). Both the angle between the right upper lobe (RUL) bronchus origin and the RMSB and the length of the RMSB can be measured with high resolution CT-scan. These measures can be useful in clinical practice as they help to determine when a R-DLT should not be used or used with caution when facing a large variation of the angle of the RUL or a proximal implantation of a RUL bronchus .

DETAILED DESCRIPTION:
Since the introduction in the early '80s of the disposable double-lumen endobronchial tube (DLT), combined with the use of fiberoptic bronchoscopy (FOB) to confirm its positioning, some controversies have aroused; the main concern being the use of the right-sided double-lumen endobronchial tube (R-DLT). Alongside this persistent controversy, the anatomy of the right tracheo-bronchial tree seems to be the principal cause of reticence for using the R-DLT. Compared to the left main stem bronchus, this anatomy is relatively complex and can be divided in two issues: 1) the variable length of the right main-stem bronchus (RMSB) and consequently, the variable level of insertion of the right upper lobe (RUL) bronchus on the lateral part of the RMSB and 2) the alignment of the lateral orifice of the R-DLT in regard of the RUL bronchus origin. A as part of an extensive study of the tracheo-bronchial tree anatomy with high resolution CT-scan, we had the opportunity to measure differently the length of the main stem right bronchus and the angulation between the RUL bronchus origin and the lateral aspect of the right side main stem bronchus.

ELIGIBILITY:
Inclusion Criteria:

* Aged 35 to 85 years old

Exclusion Criteria:

* Unavailable weight and height
* Tracheobronchial tree pathologies (e.g. : tracheomalacia, tracheobronchomegaly, endobronchial lesions, bronchiectasis, etc.)
* Mediastinal pathologies inducing an extrinsic compression of the tracheobronchial tree.
* Pulmonary pathologies inducing a deformation of the tracheobronchial tree (e.g.: retraction, important atelectasis, pulmonary fibrosis, chronic tuberculosis, etc.)
* Patients that have had a treatment or surgery inducing a deformation of the tracheobronchial tree (e.g.: lobectomy, pneumonectomy, radiotherapy)
* An important musculoskeletal deformity at the thoracic level
* Low-quality CT scan exams (e.g.: significant kinetic artifacts where measurements should be taken

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Evaluation of radiological consecutives thoracic CT-Scan reconstruction in a tertiary university hearth and lung institute. Patients had CT- scan for diagnosis or follow-up purposes
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Measurement of the length of the right mainstem bronchus | 1 day
Measure of the right upper lobe bronchus antero-posterior angulation | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Jean S. Bussières, M.D., Principal Investigator — Laval University

REFERENCES:
- [Background] McKenna MJ, Wilson RS, Botelho RJ. Right upper lobe obstruction with right-sided double-lumen endobronchial tubes: a comparison of two tube types. J Cardiothorac Anesth. 1988 Dec;2(6):734-40. doi: 10.1016/0888-6296(88)90096-8. PMID 17171882
- [Background] Klein U, Karzai W, Bloos F, Wohlfarth M, Gottschall R, Fritz H, Gugel M, Seifert A. Role of fiberoptic bronchoscopy in conjunction with the use of double-lumen tubes for thoracic anesthesia: a prospective study. Anesthesiology. 1998 Feb;88(2):346-50. doi: 10.1097/00000542-199802000-00012. PMID 9477054
- [Background] Benumof JL, Partridge BL, Salvatierra C, Keating J. Margin of safety in positioning modern double-lumen endotracheal tubes. Anesthesiology. 1987 Nov;67(5):729-38. doi: 10.1097/00000542-198711000-00018. PMID 3674473
- [Background] Benumof JL. Improving the design and function of double-lumen tubes. J Cardiothorac Anesth. 1988 Dec;2(6):729-33. doi: 10.1016/0888-6296(88)90095-6. No abstract available. PMID 17171881
- [Background] Hurford WE, Alfille PH. A quality improvement study of the placement and complications of double-lumen endobronchial tubes. J Cardiothorac Vasc Anesth. 1993 Oct;7(5):517-20. doi: 10.1016/1053-0770(93)90305-5. PMID 8268428
- [Background] Benumof JL. The position of a double-lumen tube should be routinely determined by fiberoptic bronchoscopy. J Cardiothorac Vasc Anesth. 1993 Oct;7(5):513-4. doi: 10.1016/1053-0770(93)90303-3. No abstract available. PMID 8268426
- [Background] Campos JH, Massa FC, Kernstine KH. The incidence of right upper-lobe collapse when comparing a right-sided double-lumen tube versus a modified left double-lumen tube for left-sided thoracic surgery. Anesth Analg. 2000 Mar;90(3):535-40. doi: 10.1097/00000539-200003000-00007. PMID 10702432
- [Background] Ehrenfeld JM, Walsh JL, Sandberg WS. Right- and left-sided Mallinckrodt double-lumen tubes have identical clinical performance. Anesth Analg. 2008 Jun;106(6):1847-52. doi: 10.1213/ane.0b013e31816f24d5. PMID 18499621
- [Background] Ehrenfeld JM, Mulvoy W, Sandberg WS. Performance comparison of right- and left-sided double-lumen tubes among infrequent users. J Cardiothorac Vasc Anesth. 2010 Aug;24(4):598-601. doi: 10.1053/j.jvca.2009.09.007. Epub 2009 Nov 25. PMID 19942453
- [Background] Slinger P. The clinical use of right-sided double-lumen tubes. Can J Anaesth. 2010 Apr;57(4):293-300. doi: 10.1007/s12630-009-9262-z. No abstract available. English, French. PMID 20058114
- [Background] Ikeno S, Mitsuhata H, Saito K, Hirabayashi Y, Akazawa S, Kasuda H, Shimizu R. Airway management for patients with a tracheal bronchus. Br J Anaesth. 1996 Apr;76(4):573-5. doi: 10.1093/bja/76.4.573. PMID 8652335
- [Background] Kim JH, Park SH, Han SH, Nahm FS, Jung CK, Kim KM. The distance between the carina and the distal margin of the right upper lobe orifice measured by computerised tomography as a guide to right-sided double-lumen endobronchial tube use. Anaesthesia. 2013 Jul;68(7):700-5. doi: 10.1111/anae.12208. Epub 2013 May 8. PMID 23656604
- [Background] Bussieres JS, Lacasse Y, Cote D, Beauvais M, St-Onge S, Lemieux J, Soucy J. Modified right-sided Broncho-Cath double lumen tube improves endobronchial positioning: a randomized study. Can J Anaesth. 2007 Apr;54(4):276-82. doi: 10.1007/BF03022772. PMID 17400979
- [Background] Hagihira S, Takashina M, Mashimo T. Application of a newly designed right-sided, double-lumen endobronchial tube in patients with a very short right mainstem bronchus. Anesthesiology. 2008 Sep;109(3):565-8. doi: 10.1097/ALN.0b013e31818344bd. No abstract available. PMID 18719454
- [Background] Bussieres JS, Somma J. Modified and newly designed right-sided double-lumen endobronchial tubes are complementary. Anesthesiology. 2009 May;110(5):1190; author reply 1190-1. doi: 10.1097/ALN.0b013e31819fac6a. No abstract available. PMID 19387186
- [Background] Lohser J, Umedaly HS, Fitzmaurice BG. Do-it-yourself modified right-sided Broncho-Cath double lumen tube. Can J Anaesth. 2007 Aug;54(8):675; author reply 675. doi: 10.1007/BF03022963. No abstract available. PMID 17666722
- [Background] Fischler M. A call to Mallinckrodt for a modified right-sided Broncho-Cath double lumen tube. Can J Anaesth. 2007 Dec;54(12):1029-30; author reply 1030. doi: 10.1007/BF03016642. No abstract available. PMID 18056217